CLINICAL TRIAL: NCT03536585
Title: Clinical Evaluation of the Safety and Efficacy of Using Multi-Polar RF and PEMF Technologies for the Treatment of Vaginal Laxity and for Treatment of the Mons Pubis and Labia for Improvement of Skin Laxity
Brief Title: Multi-polar RF and PEMF for Treatment of Vaginal Laxity and Mons Pubis and Labia for Improvement of Skin Laxity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CS0716
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Vulvovaginal Atrophy; Menopause; Menopause Surgical
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Independent reviewer to identify the one-month and four-month post-treatment photograph of the mons pubis and labia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vulvovaginal treatment (Experimental): Internal vaginal treatment monthly for 3 treatments; External mons pubis treatment monthly for 3 treatments; External labia treatment monthly for 3 treatments.
  Interventions: Device: Vulvovaginal treatment; Device: Baseline
- Baseline (No Intervention): Subject's baseline photograph to act as their own control for the one-month and four-month post-treatment photograph of the mons pubis and labia.

INTERVENTIONS:
Device: Vulvovaginal treatment — * Radiofrequency and pulsed electro-magnetic fields treatment of the vaginal canal to maintain an internal temperature of approximately 42 C for the proximal thermometer and 45 C for the mid and distal thermometers for 15 minutes.
  * Radiofrequency and pulsed electro-magnetic fields treatment of the labia to maintain an external temperature of approximately 40 C - 45 C for 15 minutes.
  * Radiofrequency and pulsed electro-magnetic fields treatment of the mons pubis to maintain an external temperature of approximately 40 C - 47 C for 15 minutes.
  Arms: Vulvovaginal treatment
Device: Baseline — Subject is acting as their own control. The baseline general appearance photograph will act as the comparator.
  Arms: Vulvovaginal treatment

SUMMARY:
The study evaluates the use of multi-polar radiofrequency (RF) and pulsed electro-magnetic fields (PEMF) energies for the treatment of vaginal looseness and for the treatment of the mons pubis and labia for skin tightening. All subjects will receive a total of three internal and three external treatments at four week intervals. Subjects will be followed up at one and four months after treatment is complete.

DETAILED DESCRIPTION:
Traditional non-surgical treatments to treat vaginal looseness include Kegel exercises or pelvic floor therapy with electrical stimulation of the vaginal muscles to promote muscle strength but may not be all that effective. Surgery is also used to tighten the vaginal canal and reduce the size of the mons pubis and the outer labial lips but can be associated with surgical complications. Development of new technologies to address these concerns is warranted.

Mutil-polar radiofrequency (RF) therapy to treat stress incontinence (attributed to looseness of the muscles that control the ability to hold urine) and looseness of the facial and neck skin has been used with success and minimal risk. The addition of pulsed electromagnetic field (PEMF) energy to multi-polar RF therapy has also been shown to improve the results of the RF therapy.

RF therapy has already been reported to be successful in vaginal tightening. This study will investigate whether adding PEMF to RF therapy is safe and efficacious for the treatment of vaginal loosenss. In addition, this study will also investigate whether RF and PEMF energy treatment will improve the looseness of the mons pubis and labia.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects, ≥30 years of age who are post-menopausal, or women who have undergone surgically induced menopause and are not able to bear children.
2. Requesting treatment for vaginal laxity with a score of ˂4 on the VLQ and are requesting treatment of the mons pubis and labia for skin laxity.
3. Sexual activity (vaginal intercourse minimum twice per month) in a monogamous relationship.
4. Negative Papanicolaou (Pap) Smear Cytology Test within 3 months prior to enrollment.

Exclusion Criteria:

1. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator.
2. Having a permanent implant in the treated area.
3. Prior use of collagen, fat injections and/or other methods of skin augmentation (enhancement with injected or implanted material) in the treated area within 4-6 weeks of the initial treatment or during the course of the study.
4. Use of retinoids such as oral Isotretinoin (Accutane®) within 6 months of initial treatment or during the course of the study.
5. Any other surgery in treated area within 12 months of initial treatment or during the course of the study.
6. Open laceration, abrasion or bleeding of any sort on the area to be treated.
7. Active sexual transmitted disease (STD) (e.g. genital Herpes Simplex, condylomata) or vaginosis.
8. Chronic vulvar pain or vulvar dystrophy.
9. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications, including corticosteroids, 6 months prior to and during the course of the study.
10. Having any form of active cancer at the time of enrollment and during the course of the study.
11. Significant concurrent illness, such as uncontrolled diabetes i.e. any disease state that in the opinion of the Investigator would interfere with the treatment, or healing process.
12. Having any stage 3-4 cystocele, rectocele, enterocele paravaginal defect or major pelvic organ prolapse beyond the hymenal ring.
13. Skin piercing in the treatment area.
14. Tattoos in the treatment area.
15. Prior procedure in the treated area with laser or other device within 12 months of the initial treatment or during the course of treatment.
16. History of keloid formation or poor wound healing in a previously-injured skin area.

21. History of epidermal or dermal disorders (particularly if involving collagen or microvascularity).

21. Use of an intrauterine device during the course of treatment.

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible subjects must be post-menopausal or have undergone surgical menopause.
Enrollment: 63 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Vaginal Laxity | Six months
  Self reported improvement in vaginal laxity defined as a score > 4 on Vaginal Laxity Questionnaire (VLQ) where 1 = very loose, 2 = moderately loose, 3 = slightly loose, 4 = neither tight nor loose, 5 = slightly tight, 6 = moderately tight and 7 = very tight.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Cardarelli, Study Director — Venus Concept
Locations (3):
- Canada (3):
  - Southern Health Centre, White Rock, British Columbia
  - Dr. George Arnold, Markham, Ontario
  - Pearl MD Rejuvenation, Toronto, Ontario